CLINICAL TRIAL: NCT06331286
Title: The Effect of Dulaglutide as an Adjuvant Therapy on Cognitive Function in Bipolar Disorder Patients With Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT20230091C-R1
Record Dates: First submitted 2024-03-20; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2023-08

CONDITIONS: Bipolar Disorder; Obesity; Cognition
MeSH Terms: conditions — Bipolar Disorder; Obesity | interventions — dulaglutide; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- dulaglutide injection treatment group (Experimental): 0.75mg Subcutaneous injection once a week for 24 weeks
  Interventions: Drug: dulaglutide injection
- diet and exercise guidance treatment (Other): diet and exercise guidance treatment for 24 weeks
  Interventions: Drug: dulaglutide injection

INTERVENTIONS:
Drug: dulaglutide injection — 0.75mg Subcutaneous injection once a week for 24 weeks
  Other Names: diet and exercise guidance treatment

SUMMARY:
The primary objective of this study is to investigate the effect of dulaglutide adjuvant treatment in patients with bipolar disorder with obesity, in addition to exploring the effect of GLP-1RA on cognition of bipolar disorder.

DETAILED DESCRIPTION:
3. Characteristics, composition, mechanism of action and research scope of research drugs 3.1 Dulaglutide Injection has been approved for marketing by the National Medical Products Administration (NMPA S20190022). Dulaglutide is a long-acting glucagon-like peptide-1 (GLP-1) receptor agonist with a half-life of up to 4-7 days and supports once-weekly subcutaneous administration at a dose of 0.75 mg.

The study included 60 patients (aged 18 to 65 years) with bipolar disorder with obesity who met the diagnostic criteria for bipolar disorder in the Diagnostic and Statistical Manual of Mental Disorders (DSM-5), fifth edition.Eligible patients were randomly assigned (1:1) to 24-week treatment with dulaglutide injection (n=30) or diet and exercise guidance treatment (n=30), followed up at period of enrollment as baseline and at the end of 2th, 4th，8th ，12th ，16th and 24th weeks. Adverse events were recorded.

ELIGIBILITY:
Inclusion Criteria:a. Patients (or their legal representatives/guardians) sign off-label medication and informed consent; b. 16≤ age≤ 65 years old, gender is not limited; c. Patients in the stable phase who meet the diagnostic criteria for DSM-V bipolar disorder using a short-form international neuropsychiatric interview and have kept their current medication unchanged for at least 2 months after enrollment; Body mass index (BMI) ≥28 kg/m2 ;e. Young's Mania Scale (YMRS) ≤6 points; f. HAMD-24<8 points; Han Chinese; Completed compulsory education at or above junior high school;

Exclusion Criteria:Subjects related: a. Patients who have undergone ECT therapy within 3 months; b. Have a hearing problem (inability to hear or understand the examiner's speech under normal conversation); c. Pregnant, lactating women or planning to become pregnant; d. Those who are allergic to the study drug.

Lesion-related: a. History of loss of consciousness due to cerebral organic disease or head trauma; b. Patients with any significant or unstable history of cardiovascular, respiratory, neurological (including epilepsy or significant cerebrovascular disease), renal, hepatic, or immune diseases, including inflammatory bowel disease, thyroid cancer, acute pancreatitis, etc., who are taking sulfonylurea drugs, anti-inflammatory or immunological agents, etc., especially those with a personal history or family history of medullary thyroid cancer (MTC) or 2 Patients with multiple endocrine neoplasia syndrome (MEN 2); c. Known, clinically significant laboratory markers or ECG abnormalities; Has any disease, liver disease, or renal disease that may alter the absorption, metabolism, or excretion of the study drug; d. Those with severe suicidal ideation and behavior or MARDS ≥ 30 points.

Exclusion criteria related to concomitant medications: a. chronic use of anticholinergics; b. history of psychoactive substance abuse and dependence;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
weight | Baseline, the end of Week 12 and the end of Week 24
  To analysis whether weight shows any significant trend with time changes.
Concentration of blood glucose in blood | Baseline, the end of Week 12 and the end of Week 24
  To analysis whether concentration of blood glucose in blood show any significant trend with time changes.
Concentration of total cholesterol in blood | Baseline, the end of Week 12 and the end of Week 24
  To analysis whether concentration of total cholesterol in blood show any significant trend with time changes.
Concentration of high density lipoprotein in blood | Baseline, the end of Week 12 and the end of Week 24
  To analysis whether concentration of high density lipoprotein in blood show any significant trend with time changes.
Concentration of low density lipoprotein in blood | Baseline, the end of Week 12 and the end of Week 24
  To analysis whether concentration of low density lipoprotein in blood show any significant trend with time changes.
Concentration of triglyceride in blood | Baseline, the end of Week 12 and the end of Week 24
  To analysis whether concentration of triglyceride in blood show any significant trend with time changes.
CBCT test results | Baseline, the end of Week 12 and the end of Week 24
  CBCT is a tool to measure cognitive function. It includes 4 dimensions: wire test, symbol encoding, continuous operation, and digital breadth.The wired test reflects the dimension of the speed of patient information processing. Symbolic coding reflects the patient's information processing speed, attention, working memory, reasoning, and problem-solving dimensions.
  Continuous manipulation reflects the patient's attention Dimension. The numerical breadth reflects the patient's working memory dimension.The basic information of the completion of each assessment and the completion of each assessment are calculated by the Chinese population norm model T-score, Deficit value, and extent and dimension of damage. Reflected in each assessment and the percentiles of neurocognitive function in the Chinese population.

SECONDARY OUTCOMES:
17-item Hamilton Depression Rating Scale (HAM-D17) Score | Time Frame: Baseline, the end of Week 2, 4， 8，12，16 and 24
  HAM-D17 has been the gold standard for the assessment of depression. The score needs to be based on clinical interviews, and the time frame of the assessment is usually the situation in the previous week. Most items use a 5-point scale of 0 to 4. The standard of each level is: 0 indicates none, 1 indicates mild, 2 indicates moderate, 3 indicates severe, and 4 indicates extremely severe. A few items adopt the 3-level scoring method with 0~2 points, and the grading standard is: 0 indicates none, 1 indicates mild to moderate and 2 indicates severe.
Treatment Emergent Symptom Scale (TESS) Score | Time Frame: Baseline, the end of Week 2, 4， 8，12，16 and 24
  Treatment Emergent Symptom Scale was developed by The National Institute of Mental Health (NIMH) in the USA in 1973. It is a safety assessment tool after treatment of psychiatric diseases. Evaluation is based on patient reports, physical examination results, and laboratory reports, and some items should also be consulted with the patient's family. Severity item is scored from 0 (not present) to 4 (severe). Higher scores represent a more severe condition.

CONTACTS AND LOCATIONS:
Overall Officials: Shaohua Hu, Study Director — Psychiatry, the First Affiliated Hospital, Zhejiang University School of Medicine
Locations (1):
- Department of Psychiatry, First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No